CLINICAL TRIAL: NCT00680433
Title: A Double-blind Randomised, Placebo-controlled Study of Adjunctive Ketamine Anaesthesia in ECT (Electroconvulsive Therapy)
Brief Title: Ketamine as an Anaesthetic Agent in Electroconvulsive Therapy (ECT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northside Clinic, Australia (Other)
Collaborators: Wesley Mission (Other)
Responsible Party: Principal Investigator, Colleen Loo, Associate Professor, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HREC 07281
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Major Depressive Episode
MeSH Terms: interventions — Ketamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Ketamine
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): Saline (placebo)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ketamine — Ketamine IV will be administered after the administration of the normal anaesthetic agents for ECT.
  Arms: Active
Drug: Saline — Saline (placebo) will be administered after the normal anaesthetic agents in ECT.
  Arms: Placebo

SUMMARY:
Research into the mechanisms underlying memory impairment in ECT suggests that its development may be prevented by the administration of certain medications at the time of ECT treatment. For example there are reasons to believe that ketamine, also used as an anaesthetic agent, may have such protective properties.

In this clinical study patients undergoing a course of ECT will be offered the opportunity to receive a small dose of ketamine (or a placebo) as part of their anaesthetic at the time of ECT treatment. Mood changes and any memory changes will be evaluated to see if the subjects who received ketamine had less memory side effects than those who did not, while still improving their depression.

DETAILED DESCRIPTION:
This study will report on two related trials. In the outpatient trial, patients will be administered adjunctive ketamine at two different doses (0.25mg/kg; 0.5mg/kg), and a placebo (saline), across 3 consecutive sessions within their regular maintenance ECT course. The order of conditions will be randomised across participants. Patients will be required to learn some words and faces 20 minutes prior to ECT, and complete a detailed cognitive battery 4 hours after ECT on each of the 3 occasions. The purpose of this trial is to determine whether ketamine is superior to placebo in reducing cognitive impairment following ECT and what the optimal dose of ketamine is for minimising cognitive and other side effects. Projected sample for this trial is N = 17.

In the inpatient trial, patients will be randomly assigned to receive ketamine or placebo for the duration of the acute ECT course. Patients will be administered a detailed cognitive battery the day before commencing ECT treatment, the day after the 6th treatment, and 1-3 days and 1 month following the end of the acute ECT course. The purpose of this trial is to examine whether patients in the ketamine condition had superior cognitive outcomes to those in the placebo condition during and following a course of ECT. In addition, depressive symptomatology will be examined throughout the ECT course to determine whether ketamine anaesthesia during ECT has antidepressant, as well as, cognitive benefits. Projected sample for this trial is N = 34.

This entry gives details of the main clinical trial: The effects of ketamine across a course of ECT.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy DSM-IV-TR criteria for Major Depressive Episode
* 18 years or over
* Does not have a diagnosis of schizophrenia, schizoaffective disorder, rapid cycling bipolar disorder, or current psychotic symptoms
* No known sensitivity to ketamine
* No ECT in the last 3 months
* No drug or alcohol abuse in the last 12 months
* Able to give informed consent
* Score at least 24 on Mini Mental State Examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Memory tests | Before ECT, after 6 ECT treatments, at the end of the ECT course

SECONDARY OUTCOMES:
Depression rating scale | Before ECT, after each week of treatment, at the end of the ECT course

CONTACTS AND LOCATIONS:
Overall Officials: Colleen K Loo, MB BS FRANZCP, MD, Principal Investigator — University of New South Wales
Locations (1):
- Wesley Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Background] McDaniel WW, Sahota AK, Vyas BV, Laguerta N, Hategan L, Oswald J. Ketamine appears associated with better word recall than etomidate after a course of 6 electroconvulsive therapies. J ECT. 2006 Jun;22(2):103-6. doi: 10.1097/00124509-200606000-00005. PMID 16801824
- [Background] Ostroff R, Gonzales M, Sanacora G. Antidepressant effect of ketamine during ECT. Am J Psychiatry. 2005 Jul;162(7):1385-6. doi: 10.1176/appi.ajp.162.7.1385. No abstract available. PMID 15994728
- [Background] Rasmussen KG, Jarvis MR, Zorumski CF. Ketamine anesthesia in electroconvulsive therapy. Convuls Ther. 1996 Dec;12(4):217-23. PMID 9034696
- [Background] White PF, Way WL, Trevor AJ. Ketamine--its pharmacology and therapeutic uses. Anesthesiology. 1982 Feb;56(2):119-36. doi: 10.1097/00000542-198202000-00007. No abstract available. PMID 6892475
- [Background] Krystal AD, Weiner RD, Dean MD, Lindahl VH, Tramontozzi LA 3rd, Falcone G, Coffey CE. Comparison of seizure duration, ictal EEG, and cognitive effects of ketamine and methohexital anesthesia with ECT. J Neuropsychiatry Clin Neurosci. 2003 Winter;15(1):27-34. doi: 10.1176/jnp.15.1.27. PMID 12556568
- [Background] Pigot M, Andrade C, Loo C. Pharmacological attenuation of electroconvulsive therapy--induced cognitive deficits: theoretical background and clinical findings. J ECT. 2008 Mar;24(1):57-67. doi: 10.1097/YCT.0b013e3181616c14. PMID 18379337
- [Background] MacPherson RD, Loo CK. Cognitive impairment following electroconvulsive therapy--does the choice of anesthetic agent make a difference? J ECT. 2008 Mar;24(1):52-6. doi: 10.1097/YCT.0b013e31815ef25b. PMID 18379336
- [Derived] Dean RL, Hurducas C, Hawton K, Spyridi S, Cowen PJ, Hollingsworth S, Marquardt T, Barnes A, Smith R, McShane R, Turner EH, Cipriani A. Ketamine and other glutamate receptor modulators for depression in adults with unipolar major depressive disorder. Cochrane Database Syst Rev. 2021 Sep 12;9(9):CD011612. doi: 10.1002/14651858.CD011612.pub3. PMID 34510411
- [Derived] Loo CK, Katalinic N, Garfield JB, Sainsbury K, Hadzi-Pavlovic D, Mac-Pherson R. Neuropsychological and mood effects of ketamine in electroconvulsive therapy: a randomised controlled trial. J Affect Disord. 2012 Dec 15;142(1-3):233-40. doi: 10.1016/j.jad.2012.04.032. Epub 2012 Aug 2. PMID 22858219